CLINICAL TRIAL: NCT04511039
Title: A Phase I Study of Trifluridine/ Tipiracil Plus the Poly (ADP) Ribose Polymerase Inhibitor Talazoparib in Advanced Cancers
Brief Title: Trifluridine/Tipiracil and Talazoparib for the Treatment of Patients With Locally Advanced or Metastatic Colorectal or Gastroesophageal Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: Pfizer (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 650120; R37CA282430 (NIH)
Record Dates: First submitted 2020-08-07; First posted 2020-08-12 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Advanced Malignant Solid Neoplasm; Clinical Stage III Gastroesophageal Junction Adenocarcinoma; Clinical Stage IV Gastroesophageal Junction Adenocarcinoma; Clinical Stage IVA Gastroesophageal Junction Adenocarcinoma; Clinical Stage IVB Gastroesophageal Junction Adenocarcinoma A; Locally Advanced Colorectal Carcinoma; Locally Advanced Gastroesophageal Junction Adenocarcinoma; Metastatic Colorectal Adenocarcinoma; Metastatic Gastroesophageal Junction Adenocarcinoma; Pathologic Stage III Gastroesophageal Junction Adenocarcinoma; Pathologic Stage IIIA Gastroesophageal Junction Adenocarcinoma; Pathologic Stage IIIB Gastroesophageal Junction Adenocarcinoma; Pathologic Stage IV Gastroesophageal Junction Adenocarcinoma; Pathologic Stage IVA Gastroesophageal Junction Adenocarcinoma; Pathologic Stage IVB Gastroesophageal Junction Adenocarcinoma; Postneoadjuvant Therapy Stage III Gastroesophageal Junction Adenocarcinoma AJCC v8; Postneoadjuvant Therapy Stage IIIA Gastroesophageal Junction Adenocarcinoma AJCC v8; Postneoadjuvant Therapy Stage IIIB Gastroesophageal Junction Adenocarcinoma AJCC v8; Postneoadjuvant Therapy Stage IV Gastroesophageal Junction Adenocarcinoma AJCC v8; Postneoadjuvant Therapy Stage IVA Gastroesophageal Junction Adenocarcinoma AJCC v8; Postneoadjuvant Therapy Stage IVB Gastroesophageal Junction Adenocarcinoma AJCC v8; Stage III Colorectal Cancer AJCC v8; Stage IIIA Colorectal Cancer AJCC v8; Stage IIIB Colorectal Cancer AJCC v8; Stage IIIC Colorectal Cancer AJCC v8; Stage IV Colorectal Cancer AJCC v8; Stage IVA Colorectal Cancer AJCC v8; Stage IVB Colorectal Cancer AJCC v8; Stage IVC Colorectal Cancer AJCC v8
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Trifluridine; trifluridine tipiracil drug combination; Thymidine; talazoparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): Patients receive trifluridine/tipiracil PO BID and talazoparib tosylate PO QD on days 1-5. Cycles repeat every 14 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Trifluridine and Tipiracil Hydrochloride; Drug: Talazoparib Tosylate

INTERVENTIONS:
Drug: Trifluridine and Tipiracil Hydrochloride — Given PO
  Other Names: 733030-01-8; Lonsurf; TAS 102,; Thymidine; Tipiracil Hydrochlorid Mixture with Trifluridine; Trifluridine/Tipiracil; Trifluridine/Tipiracil Hydrochloride Combination Agent TAS-102
Drug: Talazoparib Tosylate — Given PO
  Other Names: Talzenna

SUMMARY:
This phase I trial investigates the side effects and best dose of talazoparib when given together with trifluridine/tipiracil for the treatment of patients with colorectal or gastroesophageal cancer that has spread to nearby tissue or lymph nodes (locally advanced) or other places in the body (metastatic). Drugs used in the chemotherapy, such as trifluridine/tipiracil, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Talazoparib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving talazoparib with trifluridine/ tipiracil may inhibit certain enzymes in the cells that are responsible for tumor cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the safety, maximum tolerated dose (MTD), and recommended phase 2 dose (RP2D) of trifluridine and tipiracil hydrochloride (trifluridine/tipiracil [FTD/TPI]) in combination with talazoparib tosylate (talazoparib) in patients with advanced colorectal (CRC) or gastroesophageal (EGC) adenocarcinoma.

SECONDARY OBJECTIVES:

I. To determine the pharmacokinetics (PK) and pharmacodynamic (PD) markers of activity.

II. To evaluate the preliminary antineoplastic efficacy of the combination.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed CRC or EGC adenocarcinoma that is locally advanced or metastatic (Cohort A); histologically or cytologically confirmed p53mt/RASonc (Cohort B1) or p53mt/RASwt CRC (Cohort B2) that is locally advanced or metastatic. Patients with adenocarcinoma histology only are allowed to participate.
* Has received at least one prior line of therapy with progression or intolerance
* Have measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria present
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Life expectancy >= 3 months by investigator assessment
* Hemoglobin >= 9 g/dL
* Absolute neutrophil count >= 1500/mm^3
* Platelet count >= 100,000/mm^3 without transfusion or growth factor support
* Creatinine < 1.5 upper limit of normal (ULN) or creatinine clearance > 60 mL/min
* Total bilirubin < 1.5 x ULN
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 2.5 x ULN or < x 5 ULN in the presence of liver metastasis
* Albumin > 3 g/dL
* Ability to swallow oral medications
* Participants of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Systemic antineoplastic therapy within 2 weeks prior to day -14 (Dose Escalation, Cohort A) or Cycle 1 day 1 (Dose Expansion, Cohorts B1 and B2) or within the past 6 weeks if this treatment is mitomycin C or nitrosourea
* Radiotherapy within the past 2 weeks excluding palliative radiotherapy to painful bone lesions
* Prior treatment with PARP inhibitor, FUDR or FTD/TPI
* Any condition that in the investigator's opinion can limit absorption of FTD/TPI or talazoparib from the gastrointestinal (GI) tract
* Gastrointestinal obstruction (without diversion) or perforation within 4 weeks from initiation of day -14 (Dose Escalation, Cohort A) or Cycle 1 Day 1 (Dose Expansion, Cohorts B1 and B2.
* Refractory ascites (requiring weekly or more frequent paracentesis or permanent indwelling peritoneal catheter)
* Untreated central nervous system (CNS) disease. Patients with leptomeningeal disease are ineligible but patients with treated, stable CNS metastasis for at least 4 weeks are allowed to participate
* Significant cardiac disease defined as congestive heart failure stage III or IV (New York Heart Association [NYHA]), acute coronary event, cerebrovascular event, peripheral arterial embolic event, venous thromboembolic event (pulmonary embolism or lower extremity deep vein thrombosis), or ventricular arrhythmia within the past 3 months
* Other malignancy requiring active therapy
* Presence of toxicities from prior therapy of grade 2 or higher
* Active infection requiring antibiotic therapy
* Known human immunodeficiency virus (HIV) or hepatitis B infection or untreated hepatitis C infection. Patients with treated hepatitis C infection and undetectable viral load are allowed to participate
* Any history of myelodysplastic syndrome, acute leukemia, or bone marrow transplant
* Pregnant or nursing female participants
* Unwilling or unable to follow protocol requirements
* Any condition which in the investigator's opinion deems the participant an unsuitable candidate to receive study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-06-08 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events | after each cycle of treatment ( 1 cycle = 14 days)
  All adverse events will be evaluated using Common Terminology Criteria for All Adverse Events (CTCAE) version (v.) 5.
Maximum tolerated dose/ recommended phase II dose | Up to 14 days
  Will utilize the keyboard design - a novel model- assisted dose-finding method to find the maximum tolerated dose

SECONDARY OUTCOMES:
Plasma Concentration (Cmax) | Day -13 post dose
  The pharmacokinetic parameters between Trifluridine/Tipiracil and Talazoparib will be evaluated on Day -14: pre-dose, 0.5, 1, 2, 4, 6, 8 hours (hr) post-dose; day-13: 24 hr post-initial dose and day -13 pre-dose
Plasma Concentration (Cmax) | day -14 pre dose
  The pharmacokinetic parameters between Trifluridine/Tipiracil and Talazoparib will be evaluated on Day -14: pre-dose, 0.5, 1, 2, 4, 6, 8 hours (hr) post-dose; day-13: 24 hr post-initial dose and day -13 pre-dose
Plasma Concentration (Cmax) | day -14 post dose
  The pharmacokinetic parameters between Trifluridine/Tipiracil and Talazoparib will be evaluated on Day -14: pre-dose, 0.5, 1, 2, 4, 6, 8 hours (hr) post-dose; day-13: 24 hr post-initial dose and day -13 pre-dose
Plasma Concentration (Cmax) | day -13 pre dose
  The pharmacokinetic parameters between Trifluridine/Tipiracil and Talazoparib will be evaluated on Day -14: pre-dose, 0.5, 1, 2, 4, 6, 8 hours (hr) post-dose; day-13: 24 hr post-initial dose and day -13 pre-dose
Overall Response Rate (ORR) | Up to 3 years
  Will be summarized using frequencies and relative frequencies.
CEA response rate (colorectal cancer patients) | Up to 3 years
  ill be summarized using frequencies and relative frequencies. .
Progression Free Survival (PFS) | From treatment until disease progression UP to 3 years
  Will be summarized using standard Kaplan-Meier methods
Overall Survival (OS) | From treatment until death or up to 3 years
  Will be summarized using standard Kaplan-Meier methods
Progressive Disease Assessment (PD) | Up to 3 years
Number of subjects with DNA damage response | Up to 28 days prior to first drug dose, on treatment and between cylce 1-day 8 and cycle 1 day 12
  Tumor biopsies will be summarized by dose level and time-point using means and standard deviations.

CONTACTS AND LOCATIONS:
Overall Officials: Christos Fountzilas, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Yes